CLINICAL TRIAL: NCT00886782
Title: A Phase 1/2 Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BMS-863233 in Subjects With Advanced and/or Metastatic Solid Tumors
Brief Title: A Study of BMS-863233 in Patients With Advanced and/or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA198-002; EUDRACT Number: 2009-010572-20
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Cancers; Metastatic Cancer
Keywords: Advanced and/or Metastatic solid cancers
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cdc7-inhibitor (Experimental)
  Interventions: Drug: Cdc7-inhibitor

INTERVENTIONS:
Drug: Cdc7-inhibitor — Capsules, Oral, QD x 14 days until MTD is reached, 14d per 28 day cycle/QD 12 months
  Other Names: BMS-863233; XL413

SUMMARY:
The purpose of this study is to determine safety, tolerability and maximum tolerated dose of BMS-863233 in subjects advanced and/or Metastatic solid tumors.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

* Subjects with advanced and/or metastatic solid tumors who are either refractory to or have relapsed from standard therapies, or for whom a standard therapy does not exist.
* ECOG performance status ≤ 2
* Accessible for treatment, PK sample collection and required study follow-up
* Total Bilirubin ≤ 1.5 x ULN and ALT, AST ≤ 2.5 x ULN

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Subjects with known or suspected brain metastasis, primary brain tumors, or brain as the only site of disease
* Exposure to any investigational agent within 4 weeks of study drug administration
* Subjects a history of gastrointestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-05-31 (Actual); Primary Completion 2010-08-04 (Actual); Study Completion 2010-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (3):
  - Dana-Farber Cancer Institute-Vendor, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
- Canada (2):
  - Local Institution - 003, Toronto, Ontario
  - Local Institution, Toronto, Ontario
- Local Institution, Villejuif, France

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-863233 25 mg: BMS-863233 25 mg orally once daily on Days 1 to 14 of a 28-day cycle (2 weeks on treatment, 2 weeks off treatment) until progression of disease, unacceptable toxicity, withdrawal of the participant's consent, or at the discretion of the Investigator
- BMS-863233 50 mg: BMS-863233 50 mg orally once daily on Days 1 to 14 of a 28-day cycle (2 weeks on treatment, 2 weeks off treatment) until progression of disease, unacceptable toxicity, withdrawal of the participant's consent, or at the discretion of the Investigator
- BMS-863233 100 mg: BMS-863233 100 mg orally once daily on Days 1 to 14 of a 28-day cycle (2 weeks on treatment, 2 weeks off treatment) until progression of disease, unacceptable toxicity, withdrawal of the participant's consent, or at the discretion of the Investigator
Period: Overall Study
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Started | 3 | 3 | 5
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 5
Not completed — Disease progression | 3 | 3 | 3
Not completed — Study drug toxicity | 0 | 0 | 1
Not completed — Adverse event unrelated to Study drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg | Total
Number analyzed (Participants) | 3 | 3 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (14.73) | 61.0 (13.08) | 61.8 (7.60) | 60.0 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 1 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3 | 6
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 5 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) of BMS-863233
Description: DLT is defined based on adverse events that are deemed to be drug-related and occur during the first cycle of therapy using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Time Frame: Up to 28 days
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with any grade adverse events (AEs), any grade drug-related AEs, any grade serious adverse events (SAEs), any grade drug-related SAEs, and any grade AEs leading to discontinuation of any drug. The severity of AEs will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0. An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose to 30 days post last dose (Up to 14 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Participants
  AEs | 3 | 3 | 5
  Drug-related AEs | 1 | 0 | 4
  SAEs | 1 | 1 | 4
  Drug-related SAEs | 0 | 0 | 2
  AEs leading to discontinuation | 0 | 0 | 2

3. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause.
Time Frame: From first dose to 30 days post last dose (Up to 14 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Participants | 0 | 1 | 2

4. Primary Outcome: Number of Participants With Lab Abnormalities Grade 3-4
Description: Number of participants with lab abnormalities grade 3-4 including hematology, chemistry, coagulation, liver and kidney function, and electrolytes using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
  Grade 3 = severe Grade 4 = very severe
Time Frame: From first dose to 30 days post last dose (Up to 14 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Participants
  Hematology: Hemoglobin, low | 0 | 0 | 1
  Hematology: Platelet Count, low | 0 | 0 | 1
  Hematology: Lymphocytes, low | 0 | 0 | 1
  Coagulation | 0 | 0 | 0
  Liver and Kidney Function | 0 | 0 | 1
  Electrolytes: Hyponatremia, low | 1 | 0 | 1
  Electrolytes: Phosphorus, low | 0 | 0 | 1
  Other Chemistry Testing | 0 | 0 | 0

5. Secondary Outcome: BMS-863233 Maximum Observed Plasma Concentration (Cmax)
Description: BMS-863233 maximum observed plasma concentration (Cmax) is derived from plasma concentration versus time data. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: PK assessment include the following timepoints: predose, 0.5-, 1-, 2-, 4-, 5-, 6-, 8-hours end-of-infusion on Cycle 1 Day 1, Cycle 1 Day 14
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
ng/mL
  Day 1 | 904.550 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 8.638 | 2654.930 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 35.913 | 5993.514 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 50.036
  Day 14: number analyzed (Participants) | 3 | 3 | 2
  Day 14 | 907.695 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 58.219 | 1688.018 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 86.384 | 2870.897 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 37.996

6. Secondary Outcome: BMS-863233 Time of Maximum Observed Plasma Concentration (Tmax)
Description: BMS-863233 time of maximum observed plasma concentration (Tmax) is derived from plasma concentration versus time data.
Time Frame: as for outcome 5
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Hours
  Day 1 | 0.567 [0.50 to 1.00] | 0.500 [0.50 to 2.07] | 1.000 [0.50 to 2.03]
  Day 14: number analyzed (Participants) | 3 | 3 | 2
  Day 14 | 2.000 [0.63 to 2.03] | 2.000 [0.50 to 2.00] | 2.042 [2.00 to 2.08]

7. Secondary Outcome: BMS-863233 Area Under the Concentration-time Curve in One Dosing Interval (AUC(TAU))
Description: BMS-863233 Area under the concentration-time curve in one dosing interval (AUC(TAU)) is derived from plasma concentration versus time data. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: as for outcome 5
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
h*ng/mL
  Day 1 | 2317.310 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 40.781 | 8301.889 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 18.311 | 22289.734 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 63.942
  Day 14: number analyzed (Participants) | 2 | 3 | 2
  Day 14 | 2395.319 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 105.616 | 8067.026 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 57.866 | 19372.627 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 105.004

8. Secondary Outcome: BMS-863233 Clearance (CL)
Description: BMS-863233 clearance (CL) is derived from plasma concentration versus time data. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: as for outcome 5
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 2
mL/min
  Day 1: number analyzed (Participants) | 0 | 0 | 0
  Day 14 | 173.950 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 105.616 | 103.301 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 43.840 | 86.032 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 105.004

9. Secondary Outcome: BMS-863233 Effective Elimination Half-Life (T-HALFeff)
Description: Effective elimination half-life (T-HALFeff) is derived from plasma concentration versus time data.
Time Frame: PK assessment include the following timepoints: predose, 0.5-, 1-, 2-, 4-, 5-, 6-, 8-, 36-hours end-of-infusion on Cycle 1 Day 1, Cycle 1 Day 14
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 2
Hours
  Day 1: number analyzed (Participants) | 0 | 0 | 0
  Day 14 | 2.640 [1.11 to 4.17] | 4.282 [3.13 to 5.16] | 18.866 [2.31 to 35.42]

10. Secondary Outcome: BMS-863233 Accumulation Index (AI_AUC)
Description: BMS-863233 accumulation index (AI_AUC) is derived from plasma concentration versus time data. AI is calculated based on ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: as for outcome 5
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 2
Ratio
  Day 1: number analyzed (Participants) | 0 | 0 | 0
  Day 14 | 1.099 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 67.737 | 0.972 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 45.006 | 1.053 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 45.084

11. Secondary Outcome: BMS-863233 Trough Observed Plasma Concentration (Ctrough)
Description: BMS-863233 trough observed plasma concentration (Ctrough) is derived from plasma concentration versus time data. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: PK assessment include the following timepoints: predose, 0.5-, 1-, 2-, 4-, 5-, 6-, 8-, 24-hours end-of-infusion on Cycle 1 Day 2 (C1D2), (C1D7, or D8, or D9), and C1D14
Population: All participants who received at least one dose of BMS-863233 and have evaluable plasma concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 4
ng/mL
  C1D2 predose | 5.000 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 0 | 7.626 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 79.551 | 88.313 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 114.753
  C1D7, or D8, or D9 predose: number analyzed (Participants) | 0 | 3 | 3
  C1D7, or D8, or D9 predose |  | 10.068 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 47.910 | 51.789 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 166.529
  C1D14 predose: number analyzed (Participants) | 3 | 3 | 2
  C1D14 predose | 8.803 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 103.533 | 11.703 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 54.957 | 130.302 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 135.793
  C1D14 24hr postdose: number analyzed (Participants) | 3 | 3 | 3
  C1D14 24hr postdose | 8.463 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 97.338 | 14.844 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 87.332 | 34.001 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 171.563

12. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: Mean Heart Rate
Description: Baseline = Last non-missing result with a collection date-time less than the date-time of the first active dose of study medication.
Time Frame: Baseline and Predose, 2-, 4-, 8-, and 24-hours post dose on Cycle 1 Day 1 (C1D1), C3D1, C4D1, C1D2, C1D15, C3D15,
Population: All treated participants with baseline measurements
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 5
Beats/min
  2 hours post dose C1D1 | 3.5 (2.12) | 0 (7.81) | -1.4 (4.10)
  4 hours post dose C1D1: number analyzed (Participants) | 2 | 2 | 5
  4 hours post dose C1D1 | 8.0 (11.31) | 3.0 (12.73) | -1.0 (7.62)
  8 hours post dose C1D1: number analyzed (Participants) | 2 | 3 | 4
  8 hours post dose C1D1 | 7.5 (4.95) | 3.7 (5.51) | 4.3 (6.99)
  24 hours post dose C1D2: number analyzed (Participants) | 2 | 3 | 3
  24 hours post dose C1D2 | 7.5 (3.54) | -4.7 (8.33) | 1.0 (13.00)
  Predose C1D15: number analyzed (Participants) | 1 | 3 | 0
  Predose C1D15 | -2.5 (4.95) | -0.7 (5.13) |
  2 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  2 hours post dose C1D15 | 2.5 (4.95) | 0 (6.56) | 2.5 (3.54)
  4 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  4 hours post dose C1D15 | 8.0 (12.73) | 5.7 (7.09) | 9.0 (2.83)
  8 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  8 hours post dose C1D15 | 11.5 (3.54) | 10.0 (8.19) | 3.5 (0.71)
  24 hours post dose C1D15 | 11.5 (2.12) | -0.7 (6.03) | 2.0 (6.82)
  2 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D1 | -2.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D1 | 3.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D1 | 12.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 3
  24 hours post dose C3D1 | -1.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  | 2.3 (5.13)
  Predose C3D15: number analyzed (Participants) | 1 | 0 | 0
  Predose C3D15 | -3.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  2 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D15 | -7.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D15 | -4.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D15 | -1.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  24 hours post dose C3D15 | -2.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C4D1: number analyzed (Participants) | 0 | 0 | 3
  24 hours post dose C4D1 |  |  | 8.3 (5.86)

13. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval
Description: as for outcome 12
Time Frame: Baseline and Predose, 2-, 4-, 8-, and 24-hours post dose on Cycle 1 Day 1 (C1D1), C1D14, C3D1, C3D15, C4D1
Population: All treated participants with baseline measurements
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 5
msec
  2 hours post dose C1D1 | 9.0 (4.24) | -11.3 (21.20) | 1.6 (4.34)
  4 hours post dose C1D1: number analyzed (Participants) | 2 | 2 | 5
  4 hours post dose C1D1 | 6.0 (11.31) | 2.0 (11.31) | 3.6 (6.99)
  8 hours post dose C1D1: number analyzed (Participants) | 2 | 3 | 4
  8 hours post dose C1D1 | 8.0 (11.31) | -2.7 (18.58) | -2.0 (8.79)
  24 hours post dose C1D2: number analyzed (Participants) | 2 | 3 | 3
  24 hours post dose C1D2 | 4.0 (8.49) | 4.0 (10.39) | 2.7 (6.11)
  Predose C1D15: number analyzed (Participants) | 1 | 3 | 0
  Predose C1D15 | 0 (0) | 1.3 (3.06) |
  2 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  2 hours post dose C1D15 | -3.0 (4.24) | 0.7 (6.11) | -2.0 (2.83)
  4 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  4 hours post dose C1D15 | 7.0 (12.73) | 3.3 (7.57) | -3.0 (1.41)
  8 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  8 hours post dose C1D15 | -1.0 (1.41) | 2.7 (12.22) | -2.0 (2.83)
  24 hours post dose C1D15 | -5.0 (1.41) | -4.7 (12.22) | -4.0 (7.21)
  2 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D1 | 4.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D1 | 8.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D1 | 0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 3
  24 hours post dose C3D1 | 18.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  | -6.7 (7.57)
  Predose C3D15: number analyzed (Participants) | 1 | 0 | 0
  Predose C3D15 | -20.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  2 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D15 | 20.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D15 | -14.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D15 | 4.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  24 hours post dose C3D15 | 8.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C4D1: number analyzed (Participants) | 0 | 0 | 3
  24 hours post dose C4D1 |  |  | -12.7 (3.06)

14. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: QRS Interval
Description: as for outcome 12
Time Frame: Baseline and Predose, 2-, 4-, 8-, and 24-hours post dose on Cycle 1 Day 1 (C1D1), C1D14, C3D1, C3D15, C4D1
Population: All treated participants with baseline measurements
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 5
msec
  2 hours post dose C1D1 | -5.0 (1.41) | 0 (0) | 3.2 (6.26)
  4 hours post dose C1D1: number analyzed (Participants) | 2 | 2 | 5
  4 hours post dose C1D1 | -2.0 (2.83) | 0 (0) | 1.6 (8.76)
  8 hours post dose C1D1: number analyzed (Participants) | 2 | 3 | 4
  8 hours post dose C1D1 | -1.0 (1.41) | 5.3 (11.02) | 0.5 (6.61)
  24 hours post dose C1D2: number analyzed (Participants) | 2 | 3 | 3
  24 hours post dose C1D2 | -2.0 (5.66) | 3.3 (4.16) | -0.7 (14.47)
  Predose C1D15: number analyzed (Participants) | 1 | 3 | 0
  Predose C1D15 | 1.0 (1.41) | 4.0 (7.21) |
  2 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  2 hours post dose C1D15 | -1.0 (1.41) | 4.7 (6.43) | -4.0 (11.31)
  4 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  4 hours post dose C1D15 | 0 (2.83) | 8.0 (6.00) | 6.0 (2.83)
  8 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  8 hours post dose C1D15 | 0 (0) | -1.3 (1.15) | 4.0 (5.66)
  24 hours post dose C1D15 | 1.0 (4.24) | 4.0 (5.29) | 3.6 (7.13)
  2 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D1 | 0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D1 | -6.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D1 | -4.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 3
  24 hours post dose C3D1 | 0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  | -13.3 (8.33)
  Predose C3D15: number analyzed (Participants) | 1 | 0 | 0
  Predose C3D15 | -6.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  2 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D15 | -2.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D15 | -4.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D15 | -6.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  24 hours post dose C3D15 | -8.0 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C4D1: number analyzed (Participants) | 0 | 0 | 3
  24 hours post dose C4D1 |  |  | -8.7 (7.02)

15. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: QTcF Interval
Description: as for outcome 12
Time Frame: Baseline and Predose, 2-, 4-, 8-, and 24-hours post dose on Cycle 1 Day 1 (C1D1), C1D14, C3D1, C3D15, C4D1
Population: All treated participants with baseline measurements
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 2 | 3 | 5
msec
  2 hours post dose C1D1 | -8.4 (3.57) | 5.8 (8.23) | -4.8 (11.62)
  4 hours post dose C1D1: number analyzed (Participants) | 2 | 2 | 5
  4 hours post dose C1D1 | -18.0 (0.68) | 2.0 (3.42) | -9.8 (7.03)
  8 hours post dose C1D1: number analyzed (Participants) | 2 | 3 | 4
  8 hours post dose C1D1 | -16.0 (10.38) | 11.9 (16.50) | -13.2 (14.26)
  24 hours post dose C1D2: number analyzed (Participants) | 2 | 3 | 3
  24 hours post dose C1D2 | -3.8 (4.47) | 3.6 (5.43) | -19.1 (10.02)
  Predose C1D15: number analyzed (Participants) | 1 | 3 | 0
  Predose C1D15 | 5.0 (0.60) | 4.2 (7.38) |
  2 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  2 hours post dose C1D15 | -16.3 (2.83) | 7.2 (8.22) | 0.6 (7.91)
  4 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  4 hours post dose C1D15 | -17.4 (3.81) | 8.1 (6.14) | 4.6 (9.45)
  8 hours post dose C1D15: number analyzed (Participants) | 2 | 3 | 2
  8 hours post dose C1D15 | -20.5 (19.44) | 3.1 (10.47) | 1.5 (1.20)
  24 hours post dose C1D15 | -16.9 (13.77) | 5.9 (13.89) | -5.6 (6.99)
  2 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D1 | 11.4 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D1 | -3.6 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D1 | 8.5 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D1: number analyzed (Participants) | 1 | 0 | 3
  24 hours post dose C3D1 | 0.4 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  | -15.4 (9.40)
  Predose C3D15: number analyzed (Participants) | 1 | 0 | 0
  Predose C3D15 | -3.1 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  2 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  2 hours post dose C3D15 | 16.7 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  4 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  4 hours post dose C3D15 | 9.9 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  8 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  8 hours post dose C3D15 | -1.7 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C3D15: number analyzed (Participants) | 1 | 0 | 0
  24 hours post dose C3D15 | 0.8 (NA) — Standard Deviation not calculable because data were only collected for 1 participant |  |
  24 hours post dose C4D1: number analyzed (Participants) | 0 | 0 | 3
  24 hours post dose C4D1 |  |  | 3.0 (4.48)

16. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the total percentage of participants whose best response is either a complete response (CR) or a partial response (PR) defined by the RECIST criteria.
  CR= Complete disappearance of all tumor lesions. PR= Decrease, relative to baseline, of 30% or greater in the sum of the longest diameter of all "target" lesions.
Time Frame: From first dose up to 14 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Perentage of participants
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Perentage of participants | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 52.2]

17. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the total percentage of participants whose best response is complete response (CR), partial response (PR), or ≥ 4 months stable disease (SD) defined by the RECIST criteria.
  CR= Complete disappearance of all tumor lesions. PR= Decrease, relative to baseline, of 30% or greater in the sum of the longest diameter of all "target" lesions.
  SD= Failure to meet criteria for complete or partial response, in the absence of progressive disease.
Time Frame: From first dose up to 14 months
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Perentage of participants
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
Number analyzed (Participants) | 3 | 3 | 5
Perentage of participants | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8] | 40.0 [5.3 to 85.3]

ADVERSE EVENTS:
Time Frame: SAEs and AEs are assessed from first dose to 30 days post last dose (Up to 14 months). Participants were assessed for all-cause mortality from their first dose to study completion (Up to 14 months).
Arm/Group | BMS-863233 25 mg | BMS-863233 50 mg | BMS-863233 100 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 2/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 4/5
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-863233 25 mg (N=3) | BMS-863233 50 mg (N=3) | BMS-863233 100 mg (N=5)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 1
LOCALISED OEDEMA (General disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-863233 25 mg (N=3) | BMS-863233 50 mg (N=3) | BMS-863233 100 mg (N=5)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 2
VISION BLURRED (Eye disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 2
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 2 | 2
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1
FAECAL INCONTINENCE (Gastrointestinal disorders) | 0 | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 0 | 4
PROCTALGIA (Gastrointestinal disorders) | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 4
FATIGUE (General disorders) | 0 | 1 | 3
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
RHINITIS (Infections and infestations) | 1 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 1
BLOOD CREATININE (Investigations) | 0 | 1 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 | 0 | 1
WEIGHT DECREASED (Investigations) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1 | 0 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 2
HEADACHE (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1
DYSURIA (Renal and urinary disorders) | 0 | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 1 | 0
PROTEINURIA (Renal and urinary disorders) | 1 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
GENERALISED ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
FLUSHING (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.